CLINICAL TRIAL: NCT06695351
Title: Pain in Subjects with High Capacity Cognitive Abilities: a Cross Sectional Study
Brief Title: Pain in Subjects with High Capacity Cognitive Abilities
Status: Not yet recruiting | Type: Observational
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Roberto Ucero Lozano, PT, PhD, PhD, PT, MSc, CHT, Universidad Europea de Madrid
Other Study IDs: GIFTEDNESS_Pain
Record Dates: First submitted 2024-10-30; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: High Cognitive Abilities; Pain; Prevalence
Keywords: high cognitive abilities; Pain; Prevalence; Kinesiophobia; Catastrophising; giftedness
MeSH Terms: conditions — Pain; Kinesiophobia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GIFTED: Patients with high cognitive abilities

SUMMARY:
In many books and website focused in high cognitive abilities talks about pain in these subjects. However, when the investigators look for in sites like pubmed there are no literature about this topic. With this study the investigators will try to know better pain experience in this population and chronic pain prevalence

DETAILED DESCRIPTION:
It's said that people with high cognitive abilities suffered pain. However, there are no scientific literature. With this study the investigators would like to know better pain experience in this population. There are two target groups include inside this population that we consider to study: Children population and adults population.

The aim of this study is to know the prevalence of chronic pain in this population and to analize the pain experience of this population and the related psychosocial variables that can modify it, like catastrophicing, kinesiophobia, anxiety, quality of life and level of physical activity,

The investigators will use a questionnaire that includes different questionnaires like TSK-11SV, PCS, STAI, SF-36 and IPAQ and many question to evaluate the demographic factor of the sample and the prevalence

The investigators will do an statistical analysis to observe the relationship and the predictors factors

ELIGIBILITY:
Inclusion Criteria:

* People with a diagnosis of high cognitive abilities

Exclusion Criteria:

* People with incapacity to answer the questionnaire
* People that's not have a good level of Spanish language

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with a diagnosis of high cognitive abilities and spanish language
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Perceived quality of life | 1 day
  Perceived quality of life was measured with the 36Item Short Form Health Survey (SF-36) scale validated in Spanish. This self-administered scale consists of 36 items in eight domains: physical functioning, limitations due to physical problems, physical pain, social role or function, mental health, limitations due to emotional problems, vitality and general perception of health.

SECONDARY OUTCOMES:
Kinesiophobia | 1 day
  The Tampa Scale of Kinesiophobia (TSK-11) was used to assess patients' fear of moving or engaging in physical activity. We used the Spanish version of this self-administered instrument, which consists of 11 items rated on a 4-point Likert scale. The total score ranges from 11 to 44, with higher values corresponding to a greater fear of being injured again by the movement. Scores of more than 27 points are considered high. The minimum detectable change of this instrument is 5.6
Catastrophising | 1 day
  Catastrophism was assessed with the Pain Catastrophizing Scale. This scale is composed of 13 items rated on a scale from 0 to 4 points (a lower score indicates lower catastrophism). The questionnaire used is validated in Spanish
Anxiety | 1 day
  Anxiety was evaluated with the validated Spanish version of the State-Trait Anxiety inventory (STAI) questionnaire. This measuring instrument has two self-assessment scales to measure two independent anxiety concepts: state and trait. Both scales have 20 items each, which are scored on a Likert scale having four possible replies (from 0 to 3). This questionnaire presents a good internal consistency in the Spanish version in anxiety/state (Cronbach's α = .90 - .93) and in anxiety/trait (Cronbach's α = .84 - .87)
Physical activity | 1 day
  The instrument used to determine participants' PA level was the IPAQ short form. Total weekly amount of PA was calculated according to the method for computation of metabolic equivalent of task (MET)minutes/week, previously established in the IPAQ instructions for analysis and data processing of the questionnaire. Then, PA level was classified as: low (<600 METmin/week), moderate ( 600 METmin/week) and high ( 3000 METmin/week), following the same guidelines. This questionnaire has acceptable validity ( = 0.30, 95% CI: 0.23-0.36) and reliability (Spearman's =0.81, 95%CI:0.79-0.82) [30]. It has also been validated in Spain (r = 0.277; p < 0.05; 75% of specificity and sensibility; k = 0.33).

OTHER OUTCOMES:
Pain | 1 day
  The perceived pain intensity was evaluated using the visual analogue scale. This scale has shown good reliability and validity for the assessment of pain intensity.18 This measuring instrument evaluates the intensity of pain on a 10 cm line (0 being "no pain" and 10 being "the worst pain"). Participants were asked to make a mark on the line to represent the average intensity of the usual joint pain they endure in the last 30 days. Similarly, they were asked to mark the maximum degree of pain they report in the last month.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided